CLINICAL TRIAL: NCT04711031
Title: Focused Lung Ultrasound: A Prospective Cohort Study in General Practice
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Julie Jepsen Strøm, MD, PhD Student, Aalborg University
Other Study IDs: 194-1
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-08

CONDITIONS: Ultrasonography; Respiratory Tract Infections; Pneumonia; General Practice
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usual care + FLUS: At index consultation, patients will receive a FLUS examination in addition to the GP's usual care of adults presenting with symptoms of an acute LRTI.
  Interventions: Other: FLUS

INTERVENTIONS:
Other: FLUS — The participating GPs use ultrasonography on a weekly basis and will use the ultrasonography device already available to them; however, the ultrasound machine system and type of transducer will be reported. The GPs will use a 14-zone FLUS scanning protocol that has previously been validated in a general practice setting. Each of the scanning zones on the patient's left side can be denoted from 1L to 7L and from 1R to 7R on the right side. Each scanning zone should be assessed using FLUS. The transducer is placed in the middle of a scanning zone making a cross sectional image of an intercostal space and the underlying pleura blades. The patients will be examined in an upright position. The GPs will be trained in the 14-zone scanning protocol during a FLUS training program prior to recruitment of patients. FLUS pathological findings are predefined, and the variables will be dichotomized into present or not present for each scanning zone.

SUMMARY:
This is a prospective cohort study that describes focused lung ultrasound (FLUS) findings in patients presenting with symptoms of an acute lower respiratory tract infection (LRTI) in general practice in Denmark.

Ten general practitioners (GPs) will perform FLUS in addition to their usual care of adults presenting with symptoms of an acute LRTI where the GP suspects a community-acquired pneumonia (CAP). Eligible patients will consecutively be invited to participate during a two months' study period until each GP has included a total of ten patients. The GPs will register information about patients including age, gender, symptoms, clinical findings, results of any point-of-care test performed, if antibiotic treatment was prescribed and they will register information on FLUS performance and findings.

ELIGIBILITY:
Inclusion Criteria (GPs):

GPs who use PoCUS (Point-of-Care Ultrasound) at least once a week in general practice or out-of-hour services.

Inclusion Criteria (Patients):

Patients aged ≥ 18 years with acute cough (< 28 days) and at least one other symptom of an acute LRTI and where the GP suspects CAP.

Exclusion Criteria (Patients):

* Previous antibiotic prescription for the current episode of acute LRTI.
* Patients not listed with the GP (no medical record available).
* The patient is not capable of understanding and signing informed consent.
* The patient does not wish to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GPs: Eligible GPs who are interested in participating will be identified through our GP network, the Facebook page for Center for General Practice at Aalborg University, the Facebook group Ultralyd i almen praksis I Danmark [Ultrasound in general practice in Denmark] and via our collaboration with the Danish Society for Ultrasound in General Practice (DAUS). Ten GPs will be selected based on demographics, experience with PoCUS, experience with FLUS, organisational aspects of the clinic and number of years as a general practitioner.
  Patients: Eligible patients will be identified when they present to general practice. Written and oral information about the study will be provided by the GP to all potential participants and if they consent to participate, they will be included.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
FLUS findings | 2022
  Description of FLUS findings in patients with symptoms of acute LRTI in general practice where the GP suspects CAP.

SECONDARY OUTCOMES:
Distribution of FLUS findings | 2022
  Distribution of FLUS findings in each of the 14 scanning zones.
FLUS image quality | 2022
  Proportion of FLUS examinations with acceptable image quality assessed by expert reviewers.
Agreement on FLUS findings | 2022
  Level of agreement between GPs and expert reviewers on FLUS findings.
Unexpected events | 2022
  Any unexpected events during the FLUS examination.
Clinical impact of FLUS | 2022
  Clinical impact of FLUS on antibiotics prescription, working diagnosis, confidence in working diagnosis, plans for treatment and visitation.
FLUS feasibility | 2022
  Number of patients where FLUS was not performed or only partially completed and the reasons for this. Number of technical breakdowns or ultrasound machine not available.
Characteristics of patients | 2022
  Characteristics of patients including age, gender, symptoms, clinical findings, results of any point-of-care test performed, if antibiotic treatment was prescribed, referral to secondary care for other imaging, examination or treatment.
Complications and hospitalisation | 2022
  Number of reported complications and hospitalisations within 28 days of follow-up. Complications included: Empyema, lung abscess, pleural effusion or sepsis.
GP follow-up initiatives | 2022
  Any GP follow-up initiatives within 28 days of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Julie J Strøm, MD, Principal Investigator — Aalborg University
Locations (1):
- Center for General Practice at Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Strom JJ, Andersen CA, Jensen MB, Thomsen JL, Laursen CB, Skaarup SH, Schultz HHL, Hansen MP. Evaluating general practitioners' focused lung ultrasound competence and findings in patients with suspected community-acquired pneumonia in general practice. Scand J Prim Health Care. 2025 Jun;43(2):359-369. doi: 10.1080/02813432.2024.2447083. Epub 2024 Dec 30. PMID 39736112